CLINICAL TRIAL: NCT04773223
Title: Comparison of Endovascular and Open Repair of Juxta- and Pararenal Abdominal Aortic Aneurysm on Short- and Long-term Clinical Outcomes
Brief Title: Comparison of Outcomes of Complex Abdominal Aortic Aneurysm Treatment
Status: Completed | Type: Observational
Sponsor: Clinical Centre of Serbia (Other)
Collaborators: Università Vita-Salute San Raffaele (Other); Helsinki University Central Hospital (Other); Dijklander Ziekenhuis (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Petar Zlatanovic, Medical Doctor, Clinical Centre of Serbia
Other Study IDs: Complex AAA surgery
Record Dates: First submitted 2021-02-20; First posted 2021-02-26 (Actual); Results first posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-02

CONDITIONS: Juxtarenal Aortic Aneurysm; Pararenal Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Open surgery group: Patients undergoing open surgery due to juxta/pararenal abdominal aortic aneurysm
  Interventions: Procedure: Open surgery and complex EVAR due to AAA
- Endovascular group: Patients undergoing some form of endovascular abdominal aortic aneurysm repair: fenestrated, chimney, etc.
  Interventions: Procedure: Open surgery and complex EVAR due to AAA

INTERVENTIONS:
Procedure: Open surgery and complex EVAR due to AAA — There will be two cohorts:
  1. Patient undergoing open surgery
  2. Patients undergoing complex endovascular repair (fenestrated, chimney, etc.)

SUMMARY:
Background: Open repair remains the gold standard for fit patients with complex AAA. In the past decade, an evolution of devices, design, components, and delivery systems expanded the application of EVAR in these challenging anatomies. Fenestrated stent-grafts are now commercially available for the repair of complex AAA in the United States and Europe. Initial reports have demonstrated a high technical success rate, low renal dysfunction rate, and low morbidity and mortality, with promising short- and long-term results. Other reports have shown excessive morbidity and mortality with fenestrated EVAR (FEVAR). Studies comparing endovascular and open repair are sparse, especially when it concerns long-term outcomes. There are till nowadays only two propensity score-matched studies, one showing worse short-term and another long-term clinical outcome for fenestrated-branched EVAR (F/BEVAR) over open surgical repair (OSR).

Aim: The aim of this study will be to compare F/BEVAR versus open AAA repair on short- and long-term clinical outcomes for the treatment of juxta- and pararenal AAA.

Methodology: This is a prospective cohort study from the four high-volume AAA repair centers: Belgrade/Serbia, Bologna/Italy, Milan/Italy, Dijklander/Netherland, Amsterdam/Netherland, and Helsinki/Finland. Data will be collected on demographics, baseline comorbidities, AAA parameters (diameter and localization), laboratory values, intra-, and postoperative data. Follow-up examinations (clinical visits and color duplex ultrasonography, CT scans) will be performed 1, 6, and 12 months after the intervention, and annually thereafter. Propensity score analysis will be performed by matching open repair patients to endovascularly treated controlling for demographics and baseline comorbidities.

Endpoints: Primary endpoints are all-cause mortality and the freedom from aortic-related reintervention. The secondary endpoint is the 30-day complication rate, especially acute kidney injury according to the RIFLE criteria.

DETAILED DESCRIPTION:
Background Endovascular abdominal aortic aneurysm repair (EVAR) has gained widespread acceptance in the treatment of patients with abdominal aortic aneurysms (AAA). Prospective randomized trials (RCTs) have demonstrated several short-term advantages over open repair such as less blood loss, operative time, hospital stay, morbidity, and mortality. The applicability of EVAR is limited by the presence of inadequate neck or involvement of the visceral arteries. Thus consequently open AAA repair is now being performed primarily for complex aortic anatomies, such as juxtarenal and pararenal aneurysms. Open repair remains the gold standard for fit patients with complex AAA. In the past decade, an evolution of devices, design, components and delivery systems expanded the application of EVAR in these challenging anatomies. Fenestrated stent-grafts are now commercially available for the repair of complex AAA in the United States and Europe. Initial reports have demonstrated a high technical success rate, low renal dysfunction rate and low morbidity and mortality with promising short- and long-term results. Other reports have shown excessive morbidity and mortality with fenestrated EVAR (FEVAR). Studies comparing endovascular and open repair are sparse, especially when it concerns long-term outcomes. There are till nowadays only two propensity score-matched studies, one showing worse short-term and another long-term clinical outcome for fenestrated-branched EVAR (F/BEVAR) over open surgical repair (OSR). Vascular surgeons are therefore left with a paucity of data to guide decision-making.

Study objectives:

1. Primary aim: Compare Kaplan-Meier freedom from aortic related reintervention and all-cause mortality rate between endovascular and open repair group Primary endpoint: Kaplan-Meier survival rate and Kaplan-Meier aortic related reintervention rate after the patient recruitment ends
2. Secondary aim: compare short term outcomes in terms of 30-day complications rate, especially acute kidney injury according to the RIFLE criteria Secondary endpoint: 30-day complications rate, especially acute kidney injury according to the RIFLE criteria

Inclusion criteria:

* All patients (over 18 years of age) with a history of juxta- and pararenal AAA repair from January 2011 to January 2021
* All management strategies will be included (endovascular and open)

Exclusion criteria:

* Patients who are pregnant
* Patients who are under 18 years of age
* Patients who have ruptured AAA
* Patients with thoracoabdominal aortic aneurysm (ThAAA)
* Patients who have a mycotic AAA
* Patients with connective tissue disorder

Sample size To ensure sufficient statistical power to answer hypothetical questions, approximately 700 subjects will be entered into the database. Aortic-related reintervention rate is the primary endpoint being used to calculate the sample size. Assuming a difference of 7% in the late reintervention rate between endovascular and open repair, 221 patients would be required in each arm to achieve a statistical power of 85% at p=0.05. With two arms (endovascular versus open), assuming a 20% rate of missing data, a total N of 550 patients is required.

Research Design

This is a prospective study including patients treated for juxta- and pararenal AAA from 2011 through 2021 treated at six different vascular surgery centers:

1. Clinic for Vascular and Endovascular Surgery, Belgrade, Serbia
2. Department of Vascular Surgery, Policlinico S. Orsola-Malpighi, Bologna, Italy
3. Department of Vascular Surgery, San Raffaele Hospital, Milan, Italy
4. Department of Vascular Surgery, Dijklander Ziekenhuis, Hoorn, Netherlands
5. Department of Vascular Surgery, Amsterdam University Hospital, Amsterdam, Netherlands
6. Department of Vascular Surgery, Helsinki Unversity Hospital, Helsinki, Finland

Procedures Involved The study does not involve any patient contact and will not impact the care that patients receive. Data regarding the patients will be compiled and analyzed to accomplish the proposed study objectives. Data collection will include demographic information, patient-related factors, and comorbidities, diagnostic imaging information, laboratory data, surgical procedure information, complications of the surgery, and outcomes.

Multi-Institutional research After the data has been collected at a participating institution, the data will be transmitted to a central analytic center located at the Clinic for Vascular and Endovascular Surgery/Clinical Center of Serbia/Medical Faculty, University of Belgrade.

Risks to Subjects As this is a prospective observational study, there is no potential for physical risks to subjects. There is a minimal risk of breach of confidentiality that could occur when patient information is collected and analyzed for the proposed study. However, appropriate measures will be taken to minimize the risk as much as possible. All information recorded will be de-identified. This study will abide by all regulations related to protecting human subjects and protected health information.

Potential Benefits to Subjects There is no direct benefit to the subjects. However, future patients with juxta- and pararenal AAA may benefit from improved care as a result of this study.

Statistics and Data Analysis Continuous variables will be described using the median and interquartile range or mean and standard deviation. Categorical variables will be described using frequencies and percentages. Group comparisons will be performed by using the Student t-test or Mann-Whitney U test, as appropriate. Categorical data will be expressed as percentages and were compared using the chi-square test or Fisher exact test. Propensity score analysis will be performed by matching endovascular to open surgery group in a 1:1 ratio controlling for demographics, baseline comorbidities, and AAA parameters. Differences will be considered statistically significant at p < 0.05. The cumulative incidences of all-cause mortality and aortic-related complications will be estimated using the Kaplan-Meier method. Differences between curves will be tested using the log-rank test. Analyses will be done with SPSS software, version 20.0 (SPSS, Chicago, IL, USA).

Conflict of Interest The investigators have no conflict of interest to report.

Funding Source There are no plans to apply for grants or additional funding. No funding is required for the completion of this study.

Publication Plan All research personnel listed on this protocol will be eligible for authorship in any resulting abstracts and publications in accordance with the qualifications outlined by the International Committee of Medical Journal Editors. The order of authors will be determined prior to manuscript development and depend on each individual's contribution to the study.

ELIGIBILITY:
Inclusion Criteria:

* All patients (over 18 years of age) with a history of juxta- and pararenal AAA repair from January 2011 to January 2022
* All management strategies will be included (endovascular and open)

Exclusion Criteria:

* Patients who are pregnant
* Patients who are under 18 years of age
* Patients who have ruptured AAA
* Patients with thoracoabdominal aortic aneurysm (ThAAA)
* Patients who have a mycotic AAA
* Patients with connective tissue disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — more than 18 year old
Study Population: All patients with juxta/pararenal abdominal aortic aneurysm (AAA) undergoing either open surgery or complex endovascular repair.
  The definition of the juxtarenal AAA will include those with a short neck (less than 1cm).
  The definition of the pararenal AAA will include those where renal arteries originate from the aneurysm itself.
Sampling Method: Probability Sample
Enrollment: 925 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Petar Zlatanovic, MD, Principal Investigator — University Clinical Centre of Serbia
Locations (1):
- Clinical Center of Serbia, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No
This will be not available freely online, but on the request.

REFERENCES:
- [Background] Tinelli G, Crea MA, de Waure C, Di Tanna GL, Becquemin JP, Sobocinski J, Snider F, Haulon S. A propensity-matched comparison of fenestrated endovascular aneurysm repair and open surgical repair of pararenal and paravisceral aortic aneurysms. J Vasc Surg. 2018 Sep;68(3):659-668. doi: 10.1016/j.jvs.2017.12.060. Epub 2018 Mar 22. PMID 29576405
- [Background] Raux M, Patel VI, Cochennec F, Mukhopadhyay S, Desgranges P, Cambria RP, Becquemin JP, LaMuraglia GM. A propensity-matched comparison of outcomes for fenestrated endovascular aneurysm repair and open surgical repair of complex abdominal aortic aneurysms. J Vasc Surg. 2014 Oct;60(4):858-63; discussion 863-4. doi: 10.1016/j.jvs.2014.04.011. Epub 2014 May 15. PMID 24835042
- [Background] Roy IN, Millen AM, Jones SM, Vallabhaneni SR, Scurr JRH, McWilliams RG, Brennan JA, Fisher RK. Long-term follow-up of fenestrated endovascular repair for juxtarenal aortic aneurysm. Br J Surg. 2017 Jul;104(8):1020-1027. doi: 10.1002/bjs.10524. Epub 2017 Apr 12. PMID 28401533
- [Background] Ferrante AM, Moscato U, Colacchio EC, Snider F. Results after elective open repair of pararenal abdominal aortic aneurysms. J Vasc Surg. 2016 Jun;63(6):1443-50. doi: 10.1016/j.jvs.2015.12.034. Epub 2016 Mar 16. PMID 26994948

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Surgery Group: Patients undergoing open surgery due to juxta/pararenal abdominal aortic aneurysm either using transperiotoneal or retroperitoneal approach
- Endovascular Group: Patients undergoing some form of endovascular abdominal aortic aneurysm repair: fenestrated EVAR (FEVAR), branched EVAR (BEVAR), or combination of both
Period: Overall Study
Arm/Group | Open Surgery Group | Endovascular Group
Started | 668 | 257
Completed | 600 | 234
Not Completed | 68 | 23

BASELINE CHARACTERISTICS:
Groups:
- Open Surgery Group: Patients undergoing open surgery due to juxta/pararenal abdominal aortic aneurysm using transperitonel or retroperitoneal approach.
- Total: Total of all reporting groups
Arm/Group | Open Surgery Group | Endovascular Group | Total
Number analyzed (Participants) | 600 | 234 | 834
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (7.1) | 73 (6.6) | 71.9 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 25 | 175
  Male | 450 | 209 | 659
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 26.9 (3.4) | 26.7 (3.7) | 26.7 (3.6)
Current smoker [Count of Participants; unit: Participants] | 170 | 89 | 259
Hypertension [Count of Participants; unit: Participants] | 480 | 210 | 690
Hyperlipidemia [Count of Participants; unit: Participants] | 413 | 144 | 557
Diabetes mellitus [Count of Participants; unit: Participants] | 142 | 45 | 187
Coronary artery disease [Count of Participants; unit: Participants] | 253 | 84 | 337
Heart failure [Count of Participants; unit: Participants] | 61 | 29 | 90
Atrila fibrillation [Count of Participants; unit: Participants] | 90 | 36 | 126
Previos stroke/transitory ischaemic attack [Count of Participants; unit: Participants] | 100 | 47 | 147
Carotid artery disease [Count of Participants; unit: Participants] | 96 | 35 | 131
Chronic obstructive pulmonary disease [Count of Participants; unit: Participants] | 277 | 88 | 365
Chronic kidney disease [Count of Participants; unit: Participants] | 167 | 62 | 229
Peripheral arterial disease [Count of Participants; unit: Participants] | 122 | 34 | 156
History of malignant disease [Count of Participants; unit: Participants] | 109 | 51 | 160

OUTCOME MEASURES:

1. Primary Outcome: Aortic Related Reintervention.
Description: In open surgery this will include patients who were reoperated due to: graft infection, graft thrombosis, pseudoaneurysm formation, secondary AAA rupture. In endovascular group reintervention will include different reasons: endoleak, migration, thrombosis, infection, fracture, secondary AAA rupture.
Time Frame: through study completion, an average of 7 year
Measure: Count of Participants; unit: Participants
Groups:
- Open Surgery Group: Patients undergoing open surgery due to juxta/pararenal abdominal aortic aneurysm through transperitoneal or retroperitoneal approach.
Arm/Group | Open Surgery Group | Endovascular Group
Number analyzed (Participants) | 600 | 234
Participants | 44 | 63

2. Primary Outcome: All-cause Mortality
Description: Any cause of mortality duing follow-up period
Time Frame: through study completion, an average of 7 year
Measure: Count of Participants; unit: Participants
Arm/Group | Open Surgery Group | Endovascular Group
Number analyzed (Participants) | 600 | 234
Participants | 256 | 91

3. Secondary Outcome: 30-day Acute Kidney Injury
Description: Acute kidney injury was defined using RIFFLE criteria.
Time Frame: 30-day acute kidney injury
Measure: Count of Participants; unit: Participants
Arm/Group | Open Surgery Group | Endovascular Group
Number analyzed (Participants) | 600 | 234
Participants | 182 | 39

ADVERSE EVENTS:
Time Frame: 84 monhts
Arm/Group | Open Surgery Group | Endovascular Group
All-Cause Mortality (participants affected / at risk) | 256/600 | 91/234
Serious Adverse Events (participants affected / at risk) | 133/600 | 51/234
Other Adverse Events (participants affected / at risk) | 0/600 | 0/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Surgery Group (N=600) | Endovascular Group (N=234)
Spinal cord ischemia (Nervous system disorders) | 3 | 8 — Spinal cord ischemia
Acute lower limb ischemia (Vascular disorders) | 18 | 8 — Acute lower limb ischemia
Srugical bleeding (General disorders) | 38 | 12 — Surgical bleeding requiring intervention
Wound dehiscence (Skin and subcutaneous tissue disorders) | 5 | 2 — Wound dehiscence
Wound infection (Infections and infestations) | 11 | 6 — Wound infection
Colonic ischaemia (Gastrointestinal disorders) | 9 | 3 — Colonic ischaemia
Acute coronary syndrome (Cardiac disorders) | 16 | 3 — Acute coronary syndrome
Stroke or transitory ischemic attack (Nervous system disorders) | 8 | 2 — Stroke or transitory ischemic attack
Deep vein thrombosis (Vascular disorders) | 11 | 2 — Deep vein thrombosis
Prolonged intubation (Respiratory, thoracic and mediastinal disorders) | 14 | 5 — Intubation lasting longer than 5 days

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT04773223/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT04773223/ICF_001.pdf